CLINICAL TRIAL: NCT02661256
Title: Effect of Nasal Continuous Positive Airway Pressure on The Pharyngeal Swallow in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WUH 14018
Record Dates: First submitted 2016-01-04; First posted 2016-01-22 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Deglutition Disorders; Respiratory Distress Syndrome In Premature Infants; Respiratory Aspiration; Newborn, Premature
Keywords: pharyngeal swallow; airway compromise; NICU
MeSH Terms: conditions — Deglutition Disorders; Respiratory Distress Syndrome In Premature Infants; Respiratory Aspiration; Premature Birth | interventions — Continuous Positive Airway Pressure; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- on NCPAP (Active Comparator): Once consented, each participant underwent a video fluoroscopic swallow study (VFSS) while NCPAP was administered via a RAM cannula® (intervention). With the NCPAP turned on each participant was fed room temperature thin liquid barium (Varibar® Thin Liquid Barium Sulfate for Suspension) from a standard bottle (60ml Similac® Volu-Feeder® with an attached Similac® Infant Nipple and Ring (standard flow), a total of 20 swallows were recorded. These swallows were termed "on NCPAP" swallows. The swallows were assessed in real time for any swallowing dysfunction.
  Interventions: Device: NCPAP; Dietary Supplement: Varibar® Thin Liquid Barium Sulfate for Suspension
- Off NCPAP (Active Comparator): Immediately following the "on NCPAP" condition, an additional 20 swallows were recorded under VFSS with the NCPAP turned off (intervention). These swallows were termed "off NCPAP" swallows.
  Interventions: Device: NCPAP; Dietary Supplement: Varibar® Thin Liquid Barium Sulfate for Suspension

INTERVENTIONS:
Device: NCPAP — Does NCPAP induce dysphagia in neonates? Each baby will be evaluated for dysphagia (using fluoroscopy) while on NCPAP and off NCPAP.
  Other Names: Continuous Positive Airway Pressure
Dietary Supplement: Varibar® Thin Liquid Barium Sulfate for Suspension — Liquid barium is used as a contrast material to allow visualization of swallowed boluses under fluoroscopy.

SUMMARY:
Oral feeding of neonates while on nasal continuous positive airway pressure (NCPAP) is a common practice in many neonatal intensive care units (NICU) all over the country. However the safety of such practice has never been established. The Investigators hypothesize that mechanoreceptors, which should perceive sensory input from the liquid bolus, may be altered by the reception of pressurized airflow provided by the NCPAP, hence increase risk of aspiration. In this study, changes in the pharyngeal phase of swallowing were identified using video fluoroscopic swallow studies (VFSS) for infants while on NCPAP as compared to off NCPAP.

DETAILED DESCRIPTION:
Preterm infants with underdeveloped lungs and term infants with cardio-respiratory illness frequently need to be placed on ventilatory assistance. Nasal Continuous Positive Airway Pressure (NCPAP) has been proven to be an effective mode of noninvasive ventilation in neonates, as it delivers positive pressure to the airway throughout the respiratory cycle. NCPAP works by improving the breathing pattern in neonates; it increases the mean airway pressure, stents the upper airway, decreases proximal airway resistance, reduces physiological dead space, optimizes lung recruitment and improves diaphragmatic function. While many infants in the Neonatal Intensive Care Units (NICUs) require NCPAP, many of their other medical and developmental needs such as initiating oral feedings need to be addressed. Oral feeding of neonates while on NCPAP is a common practice in many NICUs, however the effect of such practice on neonatal swallowing mechanism has never been investigated.

Swallowing is a complex sensorimotor function that allows infant to safely and effectively ingest liquid nutrition. The ability of an infant to successfully feed is dependent on the precise interconnection of anatomy, physiology and neurology pathways. Afferent sequences play an integral role in the infant swallowing mechanism as sensory feedback is required during all phases of swallowing to allow appropriate positioning of anatomic structures, as well as to modulate the strength, velocity, and timing of muscle contractions. Sensory information is received from various types of sensory receptors distributed throughout the oral cavity, pharynx, larynx and esophagus. Localized areas of the infant's anatomy are known to have particular types of sensory receptors that are excited by specific stimuli which elicit appropriate motor movements.

One of the most densely populated sensory receptors are the mechanoreceptors which are sensitive to touch and pressure to help decipher the shape, texture, size and temperature of the bolus about to be swallowed. The mechanoreceptors are also sensitive to the pressure and movement of air flow during breathing.

The sensations perceived by these receptors are responsible for sending afferent sensory information to the medullary region of the brainstem where they are processed by the central pattern generators (CPGs). CPGs are composed of dedicated networks of interneurons that are responsible to sequence and activate different motor neurons at specified intensities to generate motor patterns. Both the swallowing CPG and the respiratory CPG are housed within the medulla. The close proximity of these neurons allows for precise swallow and breathing coordination. A close interrelationship between the swallowing and respiratory processes is further evident as they encompass shared anatomic structures and muscular components within the pharynx, and act as physiologically and biomechanically reciprocal events.

This close interrelationship between swallowing and breathing has led to some controversy and difference in opinion among neonatologists on the decision to start oral feedings while on NCPAP. Although there is no research directly related to the effect of NCPAP on swallowing process in neonates, NCPAP has been reported to induce dilatation of the laryngeal opening in preterm infants and inhibit the swallow reflex in adults.

For preterm infants, some neonatologists advocate initiation of oral feeds at 34 weeks gestational age, even if they require NCPAP; others strictly wait for NCPAP to be discontinued before oral feeding is established, fearing that infants may have difficulty coordinating breathing and swallowing acts, resulting in airway compromise. For term infants, many propose that oral feedings can be established once physiologic stability is demonstrated, either with or without NCPAP. Such controversies exist due to lack of evidence on the effect(s) of NCPAP on swallowing safety in human neonates.

To our knowledge no studies have been completed on human infants to evaluate the effect of NCPAP on the pharyngeal swallowing mechanism. Previous studies utilizing neonatal lambs, revealed that the application of NCPAP had no deleterious effect on cardiopulmonary safety, feeding efficiency and on nutritive swallowing- breathing coordination.

This study was designed with the aim to effectively assess the effects of NCPAP on the pharyngeal swallow mechanism in human neonates. The investigators hypothesize that the presence of NCPAP will lead to alterations in the sensorimotor sequence of the pharyngeal swallowing mechanism, increasing the risk for airway compromise and aspiration. The mechanoreceptors, which perceive sensory input from the liquid bolus, may be altered by the reception of continuous stream of airflow, provided by the NCPAP.

ELIGIBILITY:
Inclusion Criteria:

* Infants in neonatal ICU requiring NCPAP and tolerating at least 50% of their total required intake by mouth from a bottle, as determined by their medical team.

Exclusion Criteria:

* Infants with other comorbidity such as upper airway anomalies, brain injury neuromuscular disease, life threatening congenital disease. Any symptomatic intercurrent acute disease e.g. infectious disease

Ages: 34 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazeeh Hanna, MD, Principal Investigator — NYU Langone Winthrop University Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 2014- August 2015. All participants were recruited from the Neonatal Intensive Care Unit (NICU) at Winthrop University Hospital, Mineola, NY.
Pre-assignment Details: Chart review- 26 preterm infants on nCPAP. Weaned off nCPAP before approaching-10. Excluded- 4 (h/o upper airway anomalies, brain injury, etc.). Eligible-12. Declined consent -5. Consented-7. Screening and VFSS completed-7. Analyzed-7. None of the enrolled participants were excluded from the trial before assignment to groups.
Groups:
- VFSS on nCPAP Then Off nCPAP: Once consented, each participant underwent a video fluoroscopic swallow study (VFSS) while NCPAP was administered via a RAM cannula® (intervention). With the NCPAP turned on each participant was fed room temperature thin liquid barium (Varibar® Thin Liquid Barium Sulfate for Suspension) from a standard bottle (60ml Similac® Volu-Feeder® with an attached Similac® Infant Nipple and Ring (standard flow), a total of 20 swallows were recorded. These swallows were termed "on NCPAP" swallows. The swallows were assessed in real time for any swallowing dysfunction.
  Immediately following the "on NCPAP" condition, an additional 20 swallows were recorded under VFSS with the NCPAP turned off (intervention). These swallows were termed "off NCPAP" swallows.
Period: Overall Study
Arm/Group | VFSS on nCPAP Then Off nCPAP
Started | 7 (Each participant went through arms in same order: on nCPAP then off nCPAP. 1 participant at a time.)
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VFSS on nCPAP Then Off nCPAP
Number analyzed (Participants) | 7
Age, Customized [Mean (Full Range); unit: weeks] — Inclusion criteria: infants with a postmenstrual age (PMA) of 34 weeks or greater
  weeks | 37 [34.1 to 40.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Winthrop University Hospital, Mineola, NY
  Participants
    United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Pharyngeal Phase Dysphagia
Description: presence of atypical or disordered movements during the pharyngeal phase of swallowing
Time Frame: <5 seconds post swallow trigger
Measure: Count of Participants; unit: Participants
Arm/Group | on NCPAP | Off NCPAP
Number analyzed (Participants) | 7 | 7
Participants | 7 | 7

2. Secondary Outcome: Tracheal Aspiration
Description: the occurrence of barium below the level of the true vocal cords
Time Frame: <5 seconds post swallow trigger
Measure: Mean (Standard Deviation); unit: percentage of aspiration
Arm/Group | on NCPAP | Off NCPAP
Number analyzed (Participants) | 7 | 7
percentage of aspiration | 33.5 (9.4) | 14.6 (7.0)

3. Secondary Outcome: Percentage of Laryngeal Length
Description: Will be measuredmeasured by deep penetration, the occurrence of barium underneath the epiglottis, in the laryngeal vestibule to the level of the vocal folds
Time Frame: <2 seconds post swallow trigger
Measure: Mean (Standard Deviation); unit: percentage of deep penetration
Arm/Group | on NCPAP | Off NCPAP
Number analyzed (Participants) | 7 | 7
percentage of deep penetration | 43.7 (15.4) | 25.3 (8.8)

4. Secondary Outcome: Silent Aspiration
Description: The occurrence of barium below the level of the vocal folds (aspiration) with no occurrence of cough (silent). This is a measure of absence of a cough during aspiration (silent aspiration).
Time Frame: <5 seconds post swallow trigger
Measure: Count of Participants; unit: Participants
Arm/Group | on NCPAP | Off NCPAP
Number analyzed (Participants) | 7 | 7
Participants | 7 | 7

5. Secondary Outcome: Nasopharyngeal Reflux
Description: the occurrence of barium detected in the nasopharynx, posterior or superior to the velum
Time Frame: <2 seconds post swallow trigger
Measure: Mean (Standard Deviation); unit: percentage of nasopharyngeal reflux
Arm/Group | on NCPAP | Off NCPAP
Number analyzed (Participants) | 7 | 7
percentage of nasopharyngeal reflux | 42.8 (48.5) | 44.2 (45.4)

6. Secondary Outcome: Pharyngeal Residue
Description: the presence of residual barium coating the pharyngeal walls, pooling in the vallecula or pyriform sinuses post swallow (absent/mild/severe). This measure is subjective (mild = light coating and sever = significant coating of residual barium).
Time Frame: <5 seconds post swallow trigger
Measure: Number; unit: participants
Arm/Group | on NCPAP | Off NCPAP
Number analyzed (Participants) | 7 | 7
participants
  absent | 1 | 3
  mild | 4 | 4
  severe | 2 | 0

ADVERSE EVENTS:
Arm/Group | on NCPAP | Off NCPAP
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Small number of subjects: Enrollment was stopped after 7 participants due to the documented risks associated with oral feeding on NCPAP. It was unethical to expose infants to harm after clear safety risk was identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes